CLINICAL TRIAL: NCT07386522
Title: Reaching Persons With Spinal Cord Injury With Important Health Information Through a Text-messaging Intervention: Adaptation and Pilot Study
Brief Title: Health Information for Persons With Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Kerri Morgan, Associate Professor of Occupational Therapy and Neurology, Director, Research Division of Occupational Therapy, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 202402196; 1142299 (Other: Craig H. Neilsen Foundation)
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries (SCI)
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secondary Health Conditions (SHC) text message group (Active Comparator): A group provided 16-weeks of daily text messaging tips on four secondary health conditions (psychosocial health, bowel/bladder management, pressure injury/skin management, and pain).
  Interventions: Behavioral: Secondary Health Conditions (SHC) text message group
- Motivational text message group (Placebo Comparator): A group provided 16-weeks of daily motivational text messages.
  Interventions: Behavioral: Motivational text message group

INTERVENTIONS:
Behavioral: Secondary Health Conditions (SHC) text message group — The Secondary Health Conditions (SHC) text message group will participate in a 16-week text message intervention in which they will receive and respond to text messages focused on SHC information. Each domain or 4-week period will include text messages on one SHC (psychosocial health, bowel and bladder management, pressure injury/skin management, and pain). Every 4 weeks the domain topic will change until all 4 topics have been covered. On Mondays-Thursdays participants will receive messages that don't require a return response and on Fridays participants will receive a total of 5 messages, three that will require a short response. The overall goal is to provide daily tips to help manage SHC.
  Arms: Secondary Health Conditions (SHC) text message group
Behavioral: Motivational text message group — The motivational text message group will participate in a 16-week text message intervention in which the participants will receive and respond to text messages that are motivational in nature. On Mondays-Thursdays they will receive messages that don't require a return response and on Fridays participants will receive a total of 3 messages, one of those requiring a return response.
  Arms: Motivational text message group

SUMMARY:
The goal of this pilot study is to design and feasibility test a mobile phone text messaging (SMS) self-management intervention for persons with spinal cord injury (PwSCI). The project will focus on providing a 16-week text messaging intervention on the secondary health conditions of bowel/bladder management, pain, pressure injury, and psychosocial health. Our hopes are to reduce the impact of secondary health conditions (SHC) for PwSCI.

The project hopes to test whether the developed self-management program will be feasible and superior to a control group. determine the feasibility and efficacy of the SMS intervention main questions the study aims to answer are:

Participants will:

Complete an initial assessment Participate in a 16-week text messaging program using their mobile phones Complete 4-week check-ins Complete a post assessment

The main question[s] it aims to answer [is/are]:

[primary hypothesis or outcome measure 1]? [primary hypothesis or outcome measure 2]? If there is a comparison group: Researchers will compare [arm information] to see if [insert effects].

Participants will [describe the main tasks participants will be asked to do, interventions they'll be given and use bullets if it is more than 2 items].

DETAILED DESCRIPTION:
The goal of this pilot study is to build and test a mobile health (mHealth) short message service (SMS) self-management intervention for persons with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of SCI
* At least 3 months from date of injury or illness
* Identify at least one secondary health condition (pain, pressure injury, bladder/bowel dysfunction, and psychosocial distress) that impacts daily life
* Live in the community
* English as primary language
* Ability and willingness to use their own smartphone to receive and respond to text messages for the 16-week study period
* Ability and willingness to participate in two full assessments and an additional four check ins during the 16-week study period

Exclusion Criteria:

- Current admission in a hospital or in-patient rehabilitation facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
The Patient Activation Measure (PAM-13) | Baseline, every 4 weeks during 16-week intervention and up to 2 weeks post intervention
  The Patient Activation Measure (PAM-13) assesses four levels of activation: (1) the patient is disengaged and overwhelmed, (2) the patient is becoming aware but still struggling, (3) the patient takes action, and (4) the patient maintains behaviors. The psychometric properties of the PAM-13 have been assessed in multiple healthcare settings. Raw PAM-13 scores can be transformed into a continuous (0-100) scale, where higher score represent higher levels of patient activation. In order to target self-management strategies, participants will proceed through these levels.
Self-Care in Spinal Cord Injuries Inventory (SC-SCII) and Self-Care Self-Efficacy Scale in Spinal Cord Injuries (SCSES-SCI) | Baseline and up to 2 weeks post intervention
  The Self-Care in Spinal Cord Injuries Inventory and Self-Care Self-Efficacy Scale in Spinal Cord Injuries are valid and reliable instruments designed to assess self-care behaviors in individuals with spinal cord injuries. There are four self-care dimensions: self-care maintenance, self-care monitoring, self-care management and self-care self-efficacy.
  Scoring uses a 5-point rating scale. Higher scores show better self-care.

SECONDARY OUTCOMES:
Spinal Cord Injury - Quality of Life Independence measurement system (SCI-QOL) | Baseline and up to 2 weeks post intervention
  The SCI-QOL is designed as a multifaceted system for measuring patient reported outcomes across a wide variety of functioning. The SCI-QOL consists of a core set of PROMIS/Neuro-QOL items that have been optimized for people with SCI. The Pain Interference (10-item), Positive Affect and Well-being (10-item), Anxiety (9-item), Resilience (8-item), Bladder Management Difficulties (8-item), Bowel Management Difficulties (9-item), and Pressure Ulcers (7-item) item banks will be the components used in this study. Each item bank is calibrated to a mean score of 50 with a standard deviation of 10, indicating normal functioning. Higher scores on the SCI-QOL reflect greater levels of the constructs being measured.
PROMIS Item Bank v.1.0 Emotional Distress and Depression (Short Form 8b) | Baseline and up to 2 weeks post intervention
  The PROMIS item bank for emotional distress - depression is a self-report measure designed to assess the extent to which patients experience depressive symptoms over the past 7 days using a 5-point Likert scale from "never (1) to "always" (5). It consists of 8 items that evaluate symptoms such as feelings of worthlessness, hopelessness, and loss of interest in activities. PROMIS instruments are scored using item-level calibrations. PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. A higher PROMIS T-score represents more of the concept being measured.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri A Morgan, PhD, Principal Investigator — Washington University School of Medicine - Program in OT
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States